CLINICAL TRIAL: NCT06495866
Title: Ultrasound Assessment of Entheseal Sites in Patients with Seronegative Spondyloarthropathy with or Without Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aalaa Ahmed El-Sayed, resident of Physical medicine, Rheumatology and Rehabilitation Department, Sohag University
Other Study IDs: Soh-Med-24-06-19MS
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-07

CONDITIONS: Spondyloarthropathy; Fibromyalgia
Keywords: Spondyloarthropathy; Fibromyalgia; Enthesitis; Ultrasound
MeSH Terms: conditions — Spondylarthropathies; Fibromyalgia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- cases of seronegative spondyloarthropathy with fibromyalgia: cases already diagnosed as seronegative spondyloarthropathy by application of ASAS classificatin criteria for axial SpA and have concomitant fibromyalgia according to 2016 ACR criteria.
  Interventions: Radiation: ultrasound
- cases of seronegative spondyloarthropathy without fibromyalgia: cases already diagnosed as seronegative spondyloarthropathy by application of ASAS classificatin criteria for axial SpA and do not match with 2016 ACR criteria for fibromyalgia.
  Interventions: Radiation: ultrasound
- controls: control individuals will be matched for sex, age, and level of schooling without history of inflammatory joint disorders or any systemic active disease.
  Interventions: Radiation: ultrasound

INTERVENTIONS:
Radiation: ultrasound — Ultrasound finding of entheseal sites of upper & lower limbs of all groups and scoring according to enthesitis scoring system

SUMMARY:
Seronegative spondyloarthropathies are a family of joint disorders that classically include ankylosing spondylitis (AS), psoriatic arthritis (PsA), inflammatory bowel disease (IBD) associated arthritis, reactive arthritis (formerly Reiter syndrome; ReA), and undifferentiated SpA. Enthesitis, or inflammation of the sites where the tendons or ligaments insert into the bone, is a key pathological finding in SpA . It is considered the hallmark and characteristic feature of spondyloarthritis (SpA). Entheses could be classified as fibrous entheses and fibrocartilaginous entheses. Regional structural damage, such as tendon injuries and bone erosions, are frequently caused by persistent enthesitis. The healing process that follows may result in the emergence of enthesophytes and, eventually, functional impairment of related anatomic structures. Imaging modalities for evaluating entheseal lesions include conventional radiology, bone scintigraphy, magnetic resonance imaging (MRI) and power Doppler (PD) ultrasound (US). US has its own unique advantage in the diagnosis of enthesitis in AS; it uses a high-frequency or ultra-high-frequency probe that effectively visualizes the internal structure of the tendon and is recognized as the gold standard for tendon involvement.

It is superior to clinical examination in the detection of peripheral enthesitis.

Manifestations of tendon enthesitis in SpA on US include a thickened tendon, hypoechoicity, local calcification and bony erosion. Abnormal blood flow in tendon entheseal sites can be detected by Power Doppler US. Fibromyalgia (FM) is a syndrome characterized by chronic musculoskeletal pain. The main symptoms of which are muscle stiffness, joint stiffness, insomnia, fatigue, mood disorders, cognitive dysfunction, anxiety, depression, general sensitivity and the inability to carry out normal daily activities [8, 9]. It can also be associated with specific diseases, such as infections, diabetes, rheumatic diseases and psychiatric or neurological disorders. Smythe and Moldofsky later developed the name "fibromyalgia" after identifying "pain points," which are areas of severe tenderness. These points are defined as areas of hyperalgesia/allodynia when a pressure of about 4 kg causes pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfill the Assessment in Spondyloarthrits International Society (ASAS) classification criteria for Axial Spondyloarthritis.
* Age above 18 years old.
* Patient cooperative and can answer questions.
* Patients who are able and willing to give written informed consent.

Exclusion Criteria:

* Other rheumatologic or collagen diseases.
* Age below 18 years and above 60 years.
* Uncooperative patients.
* Patient not able and willing to give written informed consent.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion Criteria:
  * Patients fulfill the Assessment in Spondyloarthrits International Society (ASAS) classification criteria for Axial Spondyloarthritis.
  * Age above 18 years old.
  * Patient cooperative and can answer questions.
  * Patients who are able and willing to give written informed consent.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of ultrasound detected enthesitis among both groups and controls | 12 months
  Comparison of ultrasound detected enthesitis among patients with spondyloarthropathy with secondary fibromyalgia and those with isolated spondyloarthropathy without fibromyalgia and among controls. Cases of Spondyloarthropathy will be already diagnosed using ASAS classification criteria.
  All patients will be subjected to the following:
  1. Full medical history from the patients including Demographic data (Age Sex - Marital status - Occupation - Residence), duration of disease - The treatments that patients receive.
  2. Full clinical examination and assessment including: (a) General examination and Complete rheumatological examination. (b) ASDAS. (c) Application of 2016 ACR criteria for fibromyalgia on all SpA patients to detect cases with secondary fibromyalgia.
  3. Laboratory investigations: (complete blood picture, erythrocyte sedimentation rate, C- reactive protein).
  4. Ultrasound finding of entheseal sites of upper & lower limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R Al-Agamy, MD, Study Chair — Sohag University; Ola M Mohammed, MD, Study Director — Sohag University
Locations (1):
- Sohag University hospitals, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Healy PJ, Helliwell PS. Classification of the spondyloarthropathies. Curr Opin Rheumatol. 2005 Jul;17(4):395-9. doi: 10.1097/01.bor.0000167753.01168.bd. PMID 15956834
- [Background] Kehl AS, Corr M, Weisman MH. Review: Enthesitis: New Insights Into Pathogenesis, Diagnostic Modalities, and Treatment. Arthritis Rheumatol. 2016 Feb;68(2):312-22. doi: 10.1002/art.39458. No abstract available. PMID 26473401
- [Background] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Background] D'Agostino MA, Terslev L. Imaging Evaluation of the Entheses: Ultrasonography, MRI, and Scoring of Evaluation. Rheum Dis Clin North Am. 2016 Nov;42(4):679-693. doi: 10.1016/j.rdc.2016.07.012. Epub 2016 Sep 7. PMID 27742021